CLINICAL TRIAL: NCT03796520
Title: Clinical Validation Study of the Simplified Seizure Classification Algorithm
Brief Title: Validation Study of the Simplified Seizure Classification Algorithm
Acronym: VASSCA
Status: Completed | Type: Observational
Sponsor: Sándor Beniczky (Other)
Collaborators: Danish Epilepsy Centre (Unknown); Shiraz University of Medical Sciences (Other); University of Pavia (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: EpiPick-1
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected for epilepsy: The cohort includes patients referred to the participating centers on suspicion of epilepsy, provided their seizure onset was at 10 years of age or older.
  Interventions: Diagnostic Test: EpiPick simplified seizure classification algorithm

INTERVENTIONS:
Diagnostic Test: EpiPick simplified seizure classification algorithm — EpiPick simplified seizure classification algorithm input:
  Grey matter brain lesion Exclusively nocturnal seizures First seizure at age > 20 years Lip smacking or chewing during seizures Staring with impaired awareness, lasting less than 20s without postictal confusion Sudden irregular jerks, in isolation or brief series, if none of the following applies: Are the jerks consistently in the same limb? When resting in bed when falling asleep? Bilateral tonic-clonic seizures within 1h of awakening or immediately preceded by irregular jerks Any of the following is present: Skin turning pale pre-ictally; Loss of consciousness immediately after urination or defecation; Sudden slump with loss of awareness, lasting less than 10 seconds; Seizure lasting longer than 10 minutes, with eyes closed throughout the seizure; Severe pre-ictal headache; Episodes consisting of falls that occur always after change in posture to the upright position, or coughing or feeling pain.

SUMMARY:
An algorithm has been developed for simplified classification of epileptic seizures, in order to optimize choice of antiepileptic drugs.

The objective of this study was to clinically validate the algorithm.

DETAILED DESCRIPTION:
Optimal choice of antiepileptic drugs (AEDs) depend on the patients´ seizure-types. Over the last four decades, several classification systems have been proposed for epileptic seizures. The recent position paper of the International League Against Epilepsy defines 63 seizure-types. While this complex system might be useful for detailed phenotyping, currently there is no evidence that each of these seizure-types needs different clinical management strategy, and many clinicians find it difficult to implement.

To help physicians with optimizing the choice of AEDs, the investigators developed a simplified seizure classification, consisting of the minimal number of seizure-types, necessary for choice of AEDs, and the investigators developed an algorithm that identifies the patient´s seizure-type, based on a set of 10 simple questions, that can be answered by physicians even without extensive training in epilepsy. The current form of the algorithm was developed for patients whose seizures started in adolescence or adulthood (at the age of 10 years or older).

In this study, the investigators aim to validate the diagnostic algorithm, by comparing the seizure-type identified by the algorithm with the diagnosis and seizure-type as defined by trained experts, in the clinical workup of the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the participating centers on suspicion of epilepsy

Exclusion Criteria:

* none

Ages: 10 Years to 120 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients referred to the participating centers on suspicion of epilepsy, provided their seizure onset was at 10 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-06-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
AC1 | Through study completion, an average of 8 months.
  Agreement coefficient between index test (EpiPick) and the reference standard (expert classification)

CONTACTS AND LOCATIONS:
Overall Officials: Sandor Beniczky, MD, PhD, Principal Investigator — Aarhus University Hospital; Guido Rubboli, MD, PhD, Principal Investigator — Danich Epilepsy Centre; Michael Sperling, MD, PhD, Principal Investigator — Thomas Jefferson University; Emilio Perucca, MD, PhD, Principal Investigator — University of Pavia; Ali A Asadi-Pooya, MD, PhD, Principal Investigator — Shiraz University of Medical Sciences
Locations (5):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Danish Epilepsy Centre, Dianalund
- Shiraz University of Medical Sciences, Shiraz, Iran
- University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Age, gender, EpiPick diagnostic score, EpiPick seizure classification, reference standard, result of EEG, result of MRI.
Supporting Information: Study Protocol, SAP
Time Frame: After publication.

REFERENCES:
- [Background] Fisher RS, Cross JH, French JA, Higurashi N, Hirsch E, Jansen FE, Lagae L, Moshe SL, Peltola J, Roulet Perez E, Scheffer IE, Zuberi SM. Operational classification of seizure types by the International League Against Epilepsy: Position Paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):522-530. doi: 10.1111/epi.13670. Epub 2017 Mar 8. PMID 28276060
- [Background] Brodie MJ. Practical Use of Newer Antiepileptic Drugs as Adjunctive Therapy in Focal Epilepsy. CNS Drugs. 2015 Nov;29(11):893-904. doi: 10.1007/s40263-015-0285-4. PMID 26507832
- [Background] Brodie MJ, Covanis A, Gil-Nagel A, Lerche H, Perucca E, Sills GJ, White HS. Antiepileptic drug therapy: does mechanism of action matter? Epilepsy Behav. 2011 Aug;21(4):331-41. doi: 10.1016/j.yebeh.2011.05.025. Epub 2011 Jul 16. PMID 21763207
- [Background] Stephen LJ, Brodie MJ. Selection of antiepileptic drugs in adults. Neurol Clin. 2009 Nov;27(4):967-992. doi: 10.1016/j.ncl.2009.06.007. PMID 19853218
- [Background] Brodie MJ, Elder AT, Kwan P. Epilepsy in later life. Lancet Neurol. 2009 Nov;8(11):1019-30. doi: 10.1016/S1474-4422(09)70240-6. Epub 2009 Oct 1. PMID 19800848
- [Background] Beniczky S, Rubboli G, Aurlien H, Hirsch LJ, Trinka E, Schomer DL; SCORE consortium. The new ILAE seizure classification: 63 seizure types? Epilepsia. 2017 Jul;58(7):1298-1300. doi: 10.1111/epi.13799. No abstract available. PMID 28677857
- [Derived] Beniczky S, Asadi-Pooya AA, Perucca E, Rubboli G, Tartara E, Meritam Larsen P, Ebrahimi S, Farzinmehr S, Rampp S, Sperling MR. A web-based algorithm to rapidly classify seizures for the purpose of drug selection. Epilepsia. 2021 Oct;62(10):2474-2484. doi: 10.1111/epi.17039. Epub 2021 Aug 22. PMID 34420206